CLINICAL TRIAL: NCT05201924
Title: Bedtime Routines and Health-related Outcomes in School-age Children
Brief Title: Bedtime Routines and Children's Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Han-Yi Tsai, National Taiwan University, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202007HM010
Record Dates: First submitted 2021-12-21; First posted 2022-01-21 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Myopia; Dental Caries; Sleep; Asthenopia
Keywords: Myopia; dental caries; bedtime routine; sleep
MeSH Terms: conditions — Myopia; Dental Caries; Asthenopia

STUDY DESIGN:
Intervention Model Description: An bedtime routine interventional group and a healthy lifestyle control group
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bedtime routine (Experimental): A bedtime routine intervention handbook and check list, including bedtime brushing, limited sugar consumption around bedtime, reading books instead of using screen devices before bed, setting a regular bedtime, turning off the light, and reaching a 9 to 11-hour sleep duration
  Interventions: Behavioral: Bedtime routine
- control group (Active Comparator): healthy lifestyle checklist
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Bedtime routine — a regular routine conducted around bedtime includes brush, book reading and regular bedtime
  Arms: Bedtime routine
Behavioral: Control — a healthy control checklist
  Arms: control group

SUMMARY:
In Taiwan, the prevalence of sleep problems, myopia, and dental caries in school-age children is high. Little is known regarding the implementation of oral and vision health outcomes around bedtime. A bedtime routine intervention was conducted to improve children's oral, vision and sleep health.

DETAILED DESCRIPTION:
Background: In Taiwan, the prevalence of sleep problems, myopia, and dental caries in school-age children is high. Recent studies show that there are some linkages between sleep, myopia, and dental caries; however, most of the studies were observational studies and lack of interventional studies. In addition, little is known regarding the implementation of oral and vision health outcomes around bedtime. Establishing beneficial bedtime routines is recommended for improving health-related outcomes. Brush-Book-Bed (BBB), a bedtime routine program proposed by the American Academy of Pediatrics, has been widely applied in Western countries as a bedtime guideline. Therefore, in current research, researchers will apply the concept of BBB into practice with primary caregivers with the hope to improve sleep, dental health, and vision health outcomes.

Purpose: To compare the effectiveness of a BBB intervention group to control groups in school-age children.

Method: This study is a pilot interventional study. A total of 200 first graders will be allocated to either the intervention group or the control group. Inclusion criteria include (1) sleep duration less than 9 hours or more than 11 hours (2) average bedtime later than 9:30 p.m. Exclusion criteria include (1) intellectual disability prior to pre-school age diagnosed by physicians (2) special education students (3) less than 15 school day per month (4) medications used that influence sleep (5) congenital eye diseases (6) dental emergencies. Individual permuted block randomization will be used for the assignment. Intervention includes bedtime brushing, limited sugar consumption around bedtime, reading books instead of using screen devices before bed, setting a regular bedtime, turning off the light, and reaching a 9 to 11-hour sleep duration. Researchers will send interactive reminder messages periodically to maintain participants' compliance. Sleep questionnaires include CSHQ, modified Bedtime Routine Questionnaires, a sleep diary, Pediatric Daytime Sleepiness Scale, Questionnaire, Epworth Sleepiness Scale, and The Pittsburgh Sleep Quality Index. Oral hygiene evaluation includes salivary pH value and salivary flow rate. The near vision test and refractive error are evaluated as myopia measurements. Asthenopia pictures and critical flicker fusion frequency are used to measure subjective eye fatigue. Moreover, a self-administered questionnaire related to sleep, oral hygiene, and vision health is also measured. Intervention Feasibility will be asked with open-ended questionnaires immediately after the intervention. Data analyses will be conducted using SPSS Statistics 22.0. The findings of this pilot study will provide the basis for developing a tailored bedtime routine for Taiwanese children. which can be applied in further interventional studies. In addition, outcome indicators can act as proxies, early detection if potential risks of sleep problems, and vision or oral diseases.

Estimated Result: School-age children who receive BBB intervention will have significantly better health-related outcomes than those without after the intervention, the third and sixth months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Children whose average bedtime later than 9:30 pm
2. Children who sleep less than 9 hours or more than 11 hours

Exclusion Criteria:

1. intellectual disability prior to pre-school age diagnosed by physicians
2. special education students
3. less than 15 school day per month
4. medications used that influence sleep
5. congenital eye diseases
6. dental emergencies

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
the change of bedtime activities and sleep patterns | 7 days at baseline, three month post intervention and six month post intervention
  self-administered sleep diary, including sleep patterns, screen device use 2 hours before bedtime, caffine food intake
the change of bedtime routines | baseline, three month post intervention and six month post intervention
  Bedtime routine questionnaire (Handerson & Jordan, 2010): the subscale of bedtime consistency and bedtime adaptive activities
the change of children's sleep habits | three month post intervention and six month post intervention
  Children's sleep habits questionnaire, CSHQ (Owens et al., 2000). Higher score means more disturbed sleep. The internal consistency for both the community sample was 0.68; alpha coefficients for the various subscales of the CSHQ ranged from 0.36 (Parasomnias) to 0.70 (Bedtime Resistance) for the community sample. Test-retest reliability was acceptable (range 0.62 to 0.79).
The change of caregiver's sleep quality | baseline, three month post intervention and six month post intervention
  Pittsburgh Sleep Quality Index, PSQI (Buysse et al., 1989). The global PSQI score greater than 5 yielded a diagnostic sensitivity of 89.6% and specificity of 86.5% (kappa = 0.75, p less than 0.001) in distinguishing good and poor sleepers.
The change of caregiver's daytime sleepiness | baseline, three month post intervention and six month post intervention
  Epworth Sleepiness Scale, ESS (Johns et al., 1991). The internal consistency as measured by Cronbach's alpha was 0.88. Higher scores means more daytimes sleepiness.
The change of pediatric daytime sleepiness | baseline, three month post intervention and six month post intervention
  Pediatric Daytime Sleepiness (Drake et al., 2003). Scores ranged from 0 to 32. Mean score values in the original study were 15.3 ± 6.2. Higher scores indicate greater sleepiness.

SECONDARY OUTCOMES:
the change of myopia | baseline, three month post intervention and six month post intervention
  near vision eye chart
the change of stereopsis | baseline, three month post intervention and six month post intervention
  stereo book
the change of objective Asthenopia | baseline, three month post intervention and six month post intervention
  handy flicker for critical fusion frequency test. Normal CFF ranged between 30 to 50 Hz
the change of subjective Asthnopia | baseline, three month post intervention and six month post intervention
  self-administered pictures for eye symptoms. Higher score means more eye fatigue.
the change of oral pH | baseline, three month post intervention and six month post intervention; before bedtime after brushing and rising time before brushing
  pH values was tested using MACHEREY-NAGEL pH strips.
the change of salivary flow rate | baseline, three month post intervention and six month post intervention
  Oral Schirmer's test for five minutes before bedtime after brushing and rising time before brushing
the change of health-related cognition | baseline, three month post intervention and six month post intervention
  A total of 21 questionnaires Seven questionnaire were asked for children in eye, teeth and sleep dimension to examine the effectiveness of interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Tsai, Han-Yi, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No